CLINICAL TRIAL: NCT04853524
Title: A Phase 1, Open-label Study in Healthy Participants to Investigate the Effect of Multiple-dose JNJ-56136379 on the Single-dose Pharmacokinetics of Bictegravir, Emtricitabine, and Tenofovir Alafenamide
Brief Title: A Study of JNJ-56136379 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108977; 56136379HPB1012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-56136379; bictegravir; imidazole mustard; Racivir; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bictegravir (BIC) plus Emtricitabine (FTC) plus Tenofovir Alafenamide (TAF) plus JNJ-56136379 (Experimental): Participants will receive a single oral dose of the combination of BIC plus FTC plus TAF tablet on Day 1. Multiple oral doses of JNJ-56136379 once daily on Day 6 to Day 24. A single oral dose of the combination of BIC plus FTC plus TAF tablet on Day 20.
  Interventions: Drug: JNJ-56136379; Drug: Bictegravir (BIC) plus Emtricitabine (FTC) plus Tenofovir Alafenamide (TAF)

INTERVENTIONS:
Drug: JNJ-56136379 — JNJ-56136379 tablets will be administered orally.
Drug: Bictegravir (BIC) plus Emtricitabine (FTC) plus Tenofovir Alafenamide (TAF) — A combination of BIC, FTC and TAF will be administered orally.
  Other Names: Biktarvy

SUMMARY:
The purpose of this study is to evaluate the effect of multiple-dose JNJ-56136379 on the single-dose pharmacokinetics (PK) of the combination of bictegravir (BIC), emtricitabine (FTC), tenofovir alafenamide (TAF) in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the blood biochemistry, blood coagulation, and hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Women of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and urine pregnancy test on Day -1
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeters of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* Must have a normal 12-lead electrocardiogram (ECG) at screening, including: a) predominant sinus rhythm, b) heart rate between 45 and 100 beats per minute (bpm), extremes included, c) QT interval corrected for heart rate (QTc) interval less than or equal to (<=) 450 milliseconds (ms) in male participants/ <= 470 ms in female participants (QT interval corrected according to Fridericia [QTcF]), c) QRS interval of less than (<)120 ms, and d) PR interval <=220 ms

Exclusion Criteria:

* Having donated or lost 1 or more than 1 unit of blood (500 milliliter [mL]) or had any clinically significant abnormal bleeding in the prior 60 days before the planned first administration of a study drug
* Any history of clinically significant skin disease (as judged by the investigator) such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* A history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs
* Current human immunodeficiency virus (HIV)-1 or HIV-2 infection (confirmed by antibodies) at screening
* Clinically significant history of liver disease or renal dysfunction (estimated creatinine clearance <60 milliliter per minute [mL/min]) at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Bictegravir (BIC) and Emtricitabine (FTC) | Up to Day 25
  Plasma samples will be analyzed to determine concentrations of BIC and FTC.
Plasma Concentration of Tenofovir Alafenamide (TAF) | Up to Day 20
  Plasma samples will be analyzed to determine concentrations of TAF.
Plasma Concentration of JNJ-56136379 | Up to Day 20
  Plasma samples will be analyzed to determine concentrations of JNJ-56136379.
Urine Concentration of BIC, FTC and TAF | Up to Day 22
  Urine samples will be analyzed to determine concentrations of BIC, FTC and TAF.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability of Multiple-dose JNJ-56136379 Without and With a Single dose of Combination of BIC, FTC, and TAF | Up to Day 55
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs as a Measure of Safety and Tolerability of JNJ-56136379 | Up to Day 55
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency